CLINICAL TRIAL: NCT05117164
Title: Effect of Standardised vs Local Preoperative Enteral Feeding Practice on the Incidence of NEC in Infants With Duct Dependent Lesions: a Randomised Control Trial.
Brief Title: Enteral Feeding in Infants With Duct Dependant Lesions.
Acronym: CARDIOFEED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Joanna Seliga-Siwecka, Principal investigator, Princess Anna Mazowiecka Hospital, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CARDIOFEED
Record Dates: First submitted 2021-10-31; First posted 2021-11-11 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Duct Dependent Lesions; Necrotising Enterocolitis; Death; Growth
Keywords: congenital heart disease; nutrition; growth; newborn
MeSH Terms: conditions — Enterocolitis, Necrotizing; Death; Heart Defects, Congenital | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients will receive enteral feeding based on the practice of the leading physician.
- intervention (Experimental): Infants will receive enteral feeding based on the following protocol.
  Enteral nutrition Minimal enteral nutrition (MEN) will begin within 72 hours life at 10 to 20. mL/kg/day, via bolus gravity breast milk/donor human milk. MEN will not be included in the caloric goals.
  Advancements in feeding will be set at 20-30 mL/kg/day, but not more than 10ml per feeding portion to reach a goal of 150ml/kg/day, but not than 120ml/kg/day cases of fluid restriction).
  The goal will be to reach an overall daily caloric intake of minimum 100kcal/kg/d.
  Interventions: Other: enteral feeding as per predefined protocol

INTERVENTIONS:
Other: enteral feeding as per predefined protocol — Infants will receive enteral feeding based on the following protocol.
  Enteral nutrition Minimal enteral nutrition (MEN) will begin within 72 hours life at 10 to 20. mL/kg/day, via bolus gravity breast milk/donor human milk. MEN will not be included in the caloric goals.
  Advancements in feeding will be set at 20-30 mL/kg/day, but not more than 10ml per feeding portion to reach a goal of 150ml/kg/day, but not than 120ml/kg/day cases of fluid restriction).
  The goal will be to reach an overall daily caloric intake of minimum 100kcal/kg/d.
  Arms: intervention

SUMMARY:
This is a multicenter randomised controlled trial to assess whether standardised enteral feeding in newborns with duct dependenty congenital heart disease decreases the risk of necrotising enterocolitis (NEC). The investigators plan to include a total 384 infants. The study will be carried out in three level III hospitals in Poland. The primary end will be NEC and/or death. Secondary end points include weight gain, hospital length of stay, time required to reach full feeding.

ELIGIBILITY:
Inclusion criteria:

1. Duct dependent congenital heart disease
2. Term infants
3. Parental/legal guardian consent

Exclusion criteria:

1. Potential contradictions to early central feeding
2. Feeding intolerance
3. Hemodynamic instability
4. Death
5. > 50% formula based enteral feeding
6. Birth weight less than 2500g

Ages: 1 Minute to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Estimated)
Dates: Start 2022-08-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of final diagnosis of necrotizing enterocolitis (NEC). | up to two weeks life
  Number of infants diagnosed with NEC.
Proportion of death | up to two weeks life
  Death rate.

SECONDARY OUTCOMES:
growth | Number of infants with a significant median change from baseline within 12 months
  centimeters per week.
Proportion of number of interrupted feedings | final value within 4 weeks
  per day.
Final median value of Vasoactive support | within 4 weeks
  per day.
Median change from baseline of protein intake | within 4 weeks
  grams/kg
Median change from baseline of caloric intake | within 4 weeks
  kcal/kg/day
Proportion of final value of days required to reach full enteral feeding | within 4 weeks
  days
Proportion of final value of days on mechanical ventilation | within 4 weeks
  days
Proportion of final value of days required to regain birth weight | within 4 weeks
  grams
Median change from baseline of breastfeeding of > 50% | within 12 months
  per study arm
Proportion of culture proven late onset sepsis | 4 weeks
  per group

OTHER OUTCOMES:
Proportion of final value of age at transfer | 4 weeks
  months

CONTACTS AND LOCATIONS:
Overall Officials: Renata Bokiniec, MD PhD, Study Chair — Medical University of Warsaw; Joanna Seliga-Siwecka, MD PhD, Study Director — Medical University of Warsaw; Ariel Płotko, Principal Investigator — Medical University of Warsaw; Agata Wojcik-Sep, Principal Investigator — Medical University of Warsaw
Locations (2):
- Poland (2):
  - Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw
  - Princess Anna Mazowiecka Hospital, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seliga-Siwecka J, Plotko A, Wojcik-Sep A, Bokiniec R, Latka-Grot J, Zuk M, Furmanczyk K, Zielinski W, Chrzanowska M. Effect of standardized vs. local preoperative enteral feeding practice on the incidence of NEC in infants with duct dependent lesions: Protocol for a randomized control trial. Front Cardiovasc Med. 2022 Sep 8;9:893764. doi: 10.3389/fcvm.2022.893764. eCollection 2022. PMID 36158805